CLINICAL TRIAL: NCT01088659
Title: A Multicenter Randomised Study Comparing the Antiviral Efficacy of Pegylated Interferon-alfa-2a Plus Placebo vs. Pegylated Interferon-alfa-2a Plus Tenofovir for the Treatment of Chronic Delta Hepatitis
Brief Title: A Study of Pegasys (Peginterferon Alfa 2a) Alone or in Combination With Tenofovir in Patients With Chronic Hepatitis D.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML22364
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis D, Chronic
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — peginterferon alfa-2a; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: placebo
- 2 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: tenofovir

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180mcg sc weekly, 96 weeks
Drug: placebo — orally daily, 96 weeks
  Arms: 1
Drug: tenofovir — 245mg po daily, 96 weeks
  Arms: 2

SUMMARY:
This randomized, single blind study will compare the antiviral effect of Pegasys (pegylated interferon alfa-2a) plus placebo versus Pegasys plus tenofovir in patients with chronic hepatitis D. Patients will be randomized to receive 96 weeks of therapy with Pegasys (180 micrograms sc weekly) plus either placebo (orally daily) or tenofovir (245mg orally daily). Anticipated time on study treatment is 2+ years, target sample size is <50.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* chronic hepatitis D
* positive for HBsAg >/=6 months, for anti-HDV >/=3 months and for HDV-RNA at screening
* negative pregnancy test; fertile males and women of childbearing age should use two reliable forms of contraception throughout study

Exclusion Criteria:

* antiviral therapy for chronic hepatitis D within the previous 6 months
* previous therapy with pegylated interferon alfa
* treatment with conventional interferon alfa for >12 months
* hepatitis A or C, or HIV infection
* decompensated liver disease (Childs B-C)
* history or evidence of medical condition associated with chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02-16 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
proportion of patients becoming HDV-RNA negative | week 96

SECONDARY OUTCOMES:
HDV-RNA levels, HBsAg levels, HBV DNA, biochemical disease activity, liver histology | weeks 48, 96 and after 24 weeks of follow-up
Safety and tolerability: adverse events, laboratory parameters, vital signs | throughout 96 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Turkey (Türkiye) (6):
  - Ankara University Medical Facility; Hepatology Department, Ankara
  - Uni of Uludag Faculty of Medicine; I, Hastaliklari Anabilim Dali, Bursa
  - Dicle Uni Medical Faculty; Gastroenterology, Diyarbakır
  - Istanbul Uni Cerrahpasa Medical Faculty; Gastroenterolgy, Istanbul
  - Ege Uni Medical Faculty Izmir; Gastroenterology, Izmir
  - Dokuz Eylul University Medical Faculty; Infection, Izmir

REFERENCES:
- [Derived] Wedemeyer H, Yurdaydin C, Hardtke S, Caruntu FA, Curescu MG, Yalcin K, Akarca US, Gurel S, Zeuzem S, Erhardt A, Luth S, Papatheodoridis GV, Keskin O, Port K, Radu M, Celen MK, Idilman R, Weber K, Stift J, Wittkop U, Heidrich B, Mederacke I, von der Leyen H, Dienes HP, Cornberg M, Koch A, Manns MP; HIDIT-II study team. Peginterferon alfa-2a plus tenofovir disoproxil fumarate for hepatitis D (HIDIT-II): a randomised, placebo controlled, phase 2 trial. Lancet Infect Dis. 2019 Mar;19(3):275-286. doi: 10.1016/S1473-3099(18)30663-7. PMID 30833068